CLINICAL TRIAL: NCT02610777
Title: A Phase 2, Randomized, Controlled, Open-Label, Clinical Study of the Efficacy and Safety of Pevonedistat Plus Azacitidine Versus Single-Agent Azacitidine in Patients With Higher-Risk Myelodysplastic Syndromes, Chronic Myelomonocytic Leukemia and Low-Blast Acute Myelogenous Leukemia
Brief Title: An Efficacy and Safety Study of Pevonedistat Plus Azacitidine Versus Single-Agent Azacitidine in Participants With Higher-Risk Myelodysplastic Syndromes (HR MDS), Chronic Myelomonocytic Leukemia (CMML) and Low-Blast Acute Myelogenous Leukemia (AML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pevonedistat-2001; U1111-1169-6540 (Registry Identifier: WHO); 2015-000221-37 (EudraCT Number); REec-2016-2145 (Registry Identifier: REec); Pevonedistat-2001CTID (Other: Israel)
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Results first posted 2020-09-23 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-08

CONDITIONS: Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Acute
Keywords: Drug Therapy
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Acute | interventions — Azacitidine; pevonedistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Azacitidine 75 mg/m^2 (Active Comparator): Azacitidine 75 mg/m^2, infusion, intravenously or subcutaneously, on Day 1 through Day 5, Days 8 and 9 in 28-day treatment cycles until unacceptable toxicity, relapse, transformation to AML (for participants with HR MDS or CMML), or progressive disease (for participants with low-blast AML).
  Interventions: Drug: Azacitidine
- Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2 (Experimental): Azacitidine 75 mg/m^2, infusion, intravenously or subcutaneously, on Day 1 through Day 5, Days 8 and 9 and pevonedistat 20 mg/m^2, infusion, intravenously, on Days 1, 3, and 5 in 28-day treatment cycles until unacceptable toxicity, relapse, transformation to AML (for participants with HR MDS or CMML), or progressive disease (for participants with low-blast AML).
  Interventions: Drug: Azacitidine; Drug: Pevonedistat

INTERVENTIONS:
Drug: Azacitidine — Azacitidine intravenous or subcutaneous formulation.
Drug: Pevonedistat — Pevonedistat intravenous infusion.
  Arms: Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of pevonedistat plus azacitidine versus single-agent azacitidine in participants with HR-MDS or CMML, or low-blast AML.

DETAILED DESCRIPTION:
The drug being tested in this study is called pevonedistat. Pevonedistat is being tested to treat people with MDS or CMML, or low-blast AML as a combination treatment with azacitidine. This study will look at the overall survival, event free survival and response to treatment in people who take pevonedistat and azacitidine when compared to people who take single-agent azacitidine.

The study will enroll 120 participants. Once enrolled, participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups in 28-day treatment cycles:

* Pevonedistat 20 mg/m^2 and azacitidine 75 mg/m^2 combination
* Single-agent azacitidine 75 mg/m^2

All participants will receive azacitidine via intravenous or subcutaneous route. Participants randomized to the combination arm will also receive pevonedistat intravenous infusion.

This multi-center trial will be conducted worldwide. The overall time to participate in this study is approximately 44 months. Participants will attend the end-of-treatment visit 30 days after the last dose of study drug or before the start of subsequent anti-neoplastic therapy if that occurs sooner. Participants will enter event-free survival follow-up or response follow-up (study visits every 3 months) if their disease has not transformed to AML (for participants with HR MDS or CMML) or progressed (for participants with low-blast AML), and they have not started subsequent therapy. Participants will also enter overall survival follow-up (contacted every 3 months to document subsequent therapies and survival status).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants 18 years or older.
2. Morphologically confirmed diagnosis of MDS or nonproliferative CMML (that is, with white blood cells [WBC] <20,000 per microliter [/mcL]) or low blast AML based on 1 of the following:

   French American British (FAB) Classifications:
   * Refractory anemia with excess blasts (RAEB) - defined as having 5% to 20% myeloblasts in the bone marrow.
   * CMML with 10% to 19% myeloblasts in the bone marrow and/or 5% to 19% blasts in the blood.

   OR

   WHO Classifications:
   * RAEB 1 - defined as having 5% to 9% myeloblasts in the bone marrow.
   * RAEB 2 - defined as having 10% to 19% myeloblasts in the bone marrow and/or 5% to 19% blasts in the blood.
   * CMML 2 - defined as having 10% to 19% myeloblasts in the bone marrow and/or 5% to 19% blasts in the blood.
   * CMML 1 (Although CMML 1 is defined as having <10% myeloblasts in the bone marrow and/or <5% blasts in the blood, these participants may enroll only if bone marrow blasts >=5%.
   * WHO defined AML with 20% to 30% myeloblasts in the bone marrow and <30% myeloblasts in peripheral blood who are deemed by the investigator to be appropriate for azacitidine based therapy.
3. For MDS and CMML participants, prognostic risk category, based on the Revised International Prognostic Scoring System (IPSS R), of:

   * Very high (>6 points),
   * High (>4.5 to 6 points), or
   * Intermediate (>3 to 4.5 points): a participant determined to be in the Intermediate Prognostic Risk Category is only allowable in the setting of >=5% bone marrow myeloblasts.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
5. Clinical laboratory values within the following parameters (repeat within 3 days before the first dose of study drug if laboratory values used for randomization were obtained more than 3 days before the first dose of study drug):

   * Albumin >2.7 g/dL.
   * Total bilirubin <upper limit of normal (ULN) except in participants with Gilbert's syndrome. Participants with Gilbert's syndrome may enroll if direct bilirubin <=1.5*ULN of the direct bilirubin.
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <2.5*ULN.
   * Creatinine clearance >=50 milliliter per minutes (mL/min).
   * Hb >8 g/dL. Participants may be transfused to achieve this value. Elevated indirect bilirubin due to post transfusion hemolysis is allowed.
6. For CMML participants: WBC count <20,000/mcL before administration of the first dose of study drug on Cycle 1 Day 1; participants must have been off hydroxyurea for at least 1 week prior to WBC count assessment.
7. Ability to undergo the study required bone marrow sample collection procedures.
8. Suitable venous access for the study required blood sampling (that is, including pharmacokinetic (PK) and biomarker sampling).
9. Female participants who:

   * Are postmenopausal for at least 1 year before the Screening visit , or
   * Are surgically sterile, or
   * If they are of childbearing potential, agree to practice 1 highly effective method and 1 additional effective (barrier) method of contraception at the same time, from the time of signing the informed consent through 4 months after the last dose of study drug, or
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [example, calendar, ovulation, symptothermal, postovulation methods] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together).

   Male participants, even if surgically sterilized (that is, status postvasectomy), who:
   * Agree to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug, or
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [example, calendar, ovulation, symptothermal, postovulation methods for the female partner] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together).
10. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care.

Exclusion Criteria:

1. Previous treatment with decitabine or azacitidine or other hypomethylating agent.
2. Acute promyelocytic leukemia as diagnosed by morphologic examination of bone marrow, by fluorescent in situ hybridization or cytogenetics of peripheral blood or bone marrow, or by other accepted analysis.
3. Eligible for allogenic stem cell transplantation.
4. Participants with MDS, CMML, or low blast AML, whose only site of disease is extramedullary, example, the skin.
5. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of study procedures or could limit participant expected survival to less than 6 months.
6. Treatment with any anti leukemic/anti MDS therapies (example, lenalidomide, cytarabine, anthracyclines, purine analogs) or with any investigational products within 14 days before the first dose of any study drug.
7. Known hypersensitivity to mannitol.
8. Active uncontrolled infection or severe infectious disease, such as severe pneumonia, meningitis, or septicemia.
9. Major surgery within 14 days before first dose or a scheduled surgery during study period; insertion of a venous access device (example, catheter, port) is not considered major surgery.
10. Diagnosed or treated for another malignancy within 2 years before randomization or previously diagnosed with another malignancy and have any evidence of residual disease. Participants with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone resection.
11. Life threatening illness unrelated to cancer.
12. Prothrombin time (PT) or prolongation of the activated thromboplastin time (aPTT) >1.5 ULN or active uncontrolled coagulopathy or bleeding disorder.
13. Known human immunodeficiency virus (HIV) seropositive.
14. Known hepatitis B surface antigen seropositive, or known or suspected active hepatitis C infection. Note: Participants who have isolated positive hepatitis B core antibody (that is, in the setting of negative hepatitis B surface antigen and negative hepatitis B surface antibody) must have an undetectable hepatitis B viral load.
15. Known hepatic cirrhosis or severe pre-existing hepatic impairment.
16. Known cardiopulmonary disease defined as unstable angina, clinically significant arrhythmia, congestive heart failure (New York Heart Association [NYHA] Class III or IV) and/or myocardial infarction within 6 months prior to first dose, or severe pulmonary hypertension. As an example, well controlled atrial fibrillation would not be an exclusion whereas uncontrolled atrial fibrillation would be an exclusion.
17. Treatment with strong cytochrome P450 (CYP) 3A inhibitors or inducers within 14 days before the first dose of study drug.
18. Systemic antineoplastic therapy or radiotherapy for other malignant conditions within 12 months before the first dose of any study drug, except for hydroxyurea.
19. Female participants who are lactating and breast feeding or have a positive serum pregnancy test during the Screening period or a positive urine pregnancy test on Day 1 before first dose of study drug.
20. Female participants who intend to donate eggs (ova) during the course of this study or 4 months after receiving their last dose of study drug(s).
21. Male participants who intend to donate sperm during the course of this study or 4 months after receiving their last dose of study drug(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2019-09-04 (Actual); Study Completion 2021-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Millennium Pharmaceuticals, Inc.
Locations (59):
- United States (23):
  - University of Alabama, Birmingham, Alabama
  - Greenville Health System, Little Rock, Arkansas
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Compassionate Cancer Care Medical Group Incorporated, Riverside, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Smilow Cancer Center at Yale New Haven Hospital, New Haven, Connecticut
  - University of Miami Miller School of Medicine, Miami, Florida
  - H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - San Juan Oncology Associates, Farmington, New Mexico
  - Monter Cancer Center, Lake Success, New York
  - Weill Cornell Medical College, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Cancer Care Center of South Texas, New Braunfels, Texas
  - Nebraska Cancer Specialists, The Woodlands, Texas
  - Texas Oncology - Waco, TX, Tyler, Texas
  - University of Virginia, Charlottesville, Virginia
  - Medical Oncology Associates, Spokane, Washington
  - Yakima Valley Memorial Hospital, Yakima, Washington
- Belgium (3):
  - AZ Sint-Jan AV, Bruges, West-Vlaanderen
  - Grand Hopital de Charleroi asbl, Charleroi
  - Cliniques Universitaires UCL de Mont-Godinne, Yvoir
- Bulgaria (3):
  - University Multiprofile Hospital for Active Treatment Sv Ivan Rilski EAD, Sofia
  - Specialized Hospital for Active Treatment of Haematological Diseases - Sofia, Sofia
  - University Multi-Profile Hospital for Active Treatment Dr Georgi Stranski, Sofia
- Canada (2):
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
- Czechia (2):
  - Fakultni Nemocnice Brno, Brno
  - Fakultni Nemocnice Kralovske Vinohrady, Prague
- France (3):
  - CHU de GRENOBLE, Grenoble
  - CHRU Lille, Lille
  - Hopital Saint Louis, Paris
- Germany (2):
  - Marien Hospital Akademisches Lehrkrankenhaus, Düsseldorf
  - Universitatsklinikum Ulm, Ulm
- Ireland (2):
  - Tallaght Hospital, Dublin
  - University Hospital Galway, Galway
- Israel (3):
  - Shaare Zedek Medical Center, Jerusalem
  - ZIV Medical Center, Safed
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (4):
  - Azienda Ospedaliero Universitaria Di Bologna - Policlinico S Orsola Malpighi, Bologna
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Azienda Ospedaliera Bianchi Melacrino Morelli, Reggio Calabria
  - Azienda Ospedaliero Universitaria San Giovanni Battista Di Torino, Torino
- Zuyderland Medisch Centrum, Sittard, Netherlands
- Spain (11):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Germans Trias i Pujol, Badalona
  - ICO I'Hospitalet Hospital Duran i Reynals Instituto Catalan de Oncologia de Hospitalet (ICO), Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Malaga - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Sekeres MA, Watts J, Radinoff A, Sangerman MA, Cerrano M, Lopez PF, Zeidner JF, Campelo MD, Graux C, Liesveld J, Selleslag D, Tzvetkov N, Fram RJ, Zhao D, Bell J, Friedlander S, Faller DV, Ades L. Randomized phase 2 trial of pevonedistat plus azacitidine versus azacitidine for higher-risk MDS/CMML or low-blast AML. Leukemia. 2021 Jul;35(7):2119-2124. doi: 10.1038/s41375-021-01125-4. Epub 2021 Jan 22. No abstract available. PMID 33483617

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 45 investigative sites in the United States [US], Canada, Belgium, Bulgaria, Czech Republic, Germany, France, Israel, Italy, Spain, and Ireland from 14 April 2016 to 23 July 2021.
Pre-assignment Details: Participants diagnosed with myelomonocytic, and myelogenous leukemia were randomized into two groups in 1:1 ratio to receive single-agent azacitidine or azacitidine + pevonedistat.
Period: Overall Study
Arm/Group | Azacitidine 75 mg/m^2 | Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2
Started | 62 | 58
Response Evaluable Population (REP) (Response Evaluable Population (REP) included all participants who received at least 1 dose of study drug, have a disease assessment at baseline, and at least 1 post baseline disease assessment.) | 53 | 55
Completed | 0 | 0
Not Completed | 62 | 58
Not completed — Lost to Follow-up | 1 | 0
Not completed — Site Terminated by Sponsor | 9 | 8
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Reason not Specified | 0 | 1
Not completed — Death | 50 | 47

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (IIT) population was defined as all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Azacitidine 75 mg/m^2 | Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2 | Total
Number analyzed (Participants) | 62 | 58 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.5 (8.87) | 71.7 (9.63) | 70.6 (9.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 16 | 37
  Male | 41 | 42 | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 55 | 52 | 107
  Unknown or Not Reported | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 54 | 52 | 106
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 3 | 3 | 6
  United States | 27 | 18 | 45
  Belgium | 5 | 5 | 10
  Bulgaria | 5 | 10 | 15
  Czech Republic | 3 | 1 | 4
  Germany | 0 | 1 | 1
  Spain | 8 | 14 | 22
  France | 1 | 1 | 2
  Ireland | 1 | 0 | 1
  Israel | 3 | 0 | 3
  Italy | 6 | 5 | 11
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 169.12 (10.857) | 168.87 (7.510) | 169.00 (9.352)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 79.19 (18.471) | 75.95 (13.716) | 77.62 (16.359)
Body Surface Area [Mean (Standard Deviation); unit: square meter (m^2)] — Body surface area was defined as [height (cm) × weight (kg)/3600]½ based on height and weight collected at baseline.
  square meter (m^2) | 1.92 (0.265) | 1.88 (0.201) | 1.90 (0.236)

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death due to any cause. Participants without documented death at the time of the analysis were censored at the date the participant was last known to be alive. The Kaplan Meier estimates was used for the analysis.
Time Frame: From date of randomization until death (up to 3 years and 5 months)
Population: ITT Population was defined as all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Azacitidine 75 mg/m^2 | Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2
Number analyzed (Participants) | 62 | 58
months | 19.0 [13.57 to 27.73] | 21.8 [18.53 to 30.88]
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2; Test type: Superiority; p = 0.464, Log Rank — P-value is from an unstratified log-rank test; Hazard Ratio (HR) = 0.861, 95% CI 2-sided [0.577 to 1.286] — Hazard Ratio (HR) was based on an unstratified Cox proportional hazard regression model with treatment as a factor

2. Secondary Outcome: Event-Free Survival (EFS)
Description: EFS is defined as the time from the date of randomization to the date of the occurrence of an event. An event is defined as death or transformation to AML for HR MDS/CMML participants, whichever occurs first, or defined as death for low-blast AML participants. HR MDS/CMML participants without documented EFS event will be censored at the date of the last response assessment. HR MDS/CMML participants with no response assessment and no death will be censored at the date of randomization. Low-blast AML participants without documentation of death will be censored at the date the participant was last known to be alive. HR MDS/CMML participants who received alternative antineoplastic therapy before death or transformation to AML will be censored at the date of last adequate assessment prior to starting alternate antineoplastic therapy. The Kaplan-Meier estimate was used for the analysis.
Time Frame: From date of randomization until transformation to AML, or death due to any cause (up to approximately 5 years)
Population: ITT Population was defined as all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Azacitidine 75 mg/m^2 | Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2
Number analyzed (Participants) | 62 | 58
months | 17.6 [11.96 to 20.50] | 21.0 [17.41 to 28.02]
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2; Event-Free Survival (EFS); Test type: Superiority; p = 0.092, Log Rank — P-value comparing EFS between treatment groups was based on the unstratified log-rank test; Hazard Ratio (HR) = 0.706, 95% CI 2-sided [0.469 to 1.061] — HR:unadjusted stratified Cox proportional hazard regression with stratification(low-blast AML,IPSS-R risk groups=very high,high,or intermediate for HRMDS/CMML),treatment as factor.HR<1:better prevention of EFS in combination arm than azacitidine arm

3. Secondary Outcome: Six-month Survival Rate
Description: Kaplan-Meier estimate of probability of OS at the end of the month 6 from randomization.
Time Frame: Month 6
Population: ITT Population was defined as all participants who were randomized. Overall number analyzed are the number of participants with data available for analyses.
Measure: Number (95% Confidence Interval); unit: survival probability
Arm/Group | Azacitidine 75 mg/m^2 | Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2
Number analyzed (Participants) | 50 | 53
survival probability | 0.806 [0.684 to 0.885] | 0.914 [0.805 to 0.963]

4. Secondary Outcome: One-year Survival Rate
Description: Kaplan-Meier estimate of probability of OS at the end of the first year from randomization.
Time Frame: Month 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: survival probability
Arm/Group | Azacitidine 75 mg/m^2 | Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2
Number analyzed (Participants) | 42 | 49
survival probability | 0.677 [0.546 to 0.778] | 0.845 [0.723 to 0.916]

5. Secondary Outcome: Time to AML Transformation in HR MDS or CMML Participants
Description: Time to AML transformation in HR MDS and CMML participants is defined as time from randomization to documented AML transformation. Participants without documented AML transformation at the time of the analysis are censored at the date of the last assessment. Participants who died before progression to AML are censored at the date of death. Transformation to AML is defined, according to World Health Organization (WHO) classification, as a participant having >20% blasts in the blood or marrow and increase of blast count by 50%.
Time Frame: From date of randomization until transformation to AML (up to approximately 5 years)
Population: ITT Population was defined as all participants who were randomized. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Azacitidine 75 mg/m^2 | Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2
Number analyzed (Participants) | 43 | 41
months | NA [NA to NA] — The median and 95% confidence interval (CI) was not estimable as participants were censored. | NA [NA to NA] — The median and 95% CI was not estimable as the participants were censored.
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2; Test type: Superiority; p = 0.267, Log Rank — P-value is from an unstratified log-rank test; Hazard Ratio (HR) = 0.562, 95% CI 2-sided [0.200 to 1.579] — Hazard ratio (HR) is based on an unstratified Cox proportional hazard regression model with treatment as a factor

6. Secondary Outcome: Percentage of Participants With Complete Remission (CR)
Description: Disease responses for HR MDS or CMML is based on the modified International Working Group (IWG) response criteria for MDS and for low-blast AML on the revised IWG response criteria for AML. CR for HR MDS or CMML: <= 5% myeloblasts with normal maturation of all cell lines in the bone marrow, and >= 11 gram/deciliter (g/dL) hemoglobin (Hb), >=100*10^9/liter (/L) platelets (plt), >=1.0*10^9/L absolute neutrophil count (ANC) and 0% blasts in peripheral blood. CR for low-blast AML: morphologic leukemia-free state, ANC of more than 1.0*10^9/L and plt of >=1.0*10^9/L, transfusion independence, and no residual evidence of extramedullary leukemia. CR with incomplete blood count recovery for low-blast AML: some participants fulfill all of the criteria for CR except for residual neutropenia (<1.0*10^9/L) or thrombocytopenia (TTP) (<100*10^9/L). The percentages are rounded off to report the nearest whole numbers.
Time Frame: From date of randomization until CR (up to approximately 5 years)
Population: Response-Evaluable Population (REP) included all participants who received at least 1 dose of study drug and had a Baseline and at least 1 postbaseline disease assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Azacitidine 75 mg/m^2 | Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2
Number analyzed (Participants) | 53 | 55
percentage of participants | 36 | 45
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2; Test type: Superiority; p = 0.312, Cochran-Mantel-Haenszel — P-value is from an unstratified Cochran-Mantel Haenszel chi-square test; Absolute Rate Difference = 9.61, 95% CI 2-sided [-8.83 to 28.04] — Absolute difference >0 represent better response achieved on pevonedistat combination compared to azacitidine treatment alone

7. Secondary Outcome: Percentage of Participants With CR and Partial Remission (PR)
Description: Disease responses for HR MDS/CMML per modified IWG response criteria for MDS and for low-blast AML on revised IWG response criteria for AML.CR for HR MDS/CMML: <=5% myeloblasts with normal maturation of all cell lines in bone marrow ,>=11 g/dL Hb;>=100*10^9/L plt; >=1.0*10^9/L ANC and 0% blasts in peripheral blood. PR for HR MDS/CMML:considered achieved if all CR criteria is met except for bone marrow blasts decreased by >=50%over pretreatment but still >5%. CR for low-blast AML: morphologic leukemia-free state, ANC of >1.0*10^9/L and plt of >=100*10^9/L, transfusion independence, no residual evidence of extramedullary leukemia. CR with incomplete blood count recovery for low-blast AML:fulfill all criteria for CR except for residual neutropenia (<100*10^9/L)/TTP(<100*10^9/L). PR for low-blast AML:all hematological values for CR but with decrease of >=50% in percentage of blasts to 5%-25% in bone marrow aspirate. The percentages are rounded off to report the nearest whole numbers.
Time Frame: From date of randomization until CR and PR (up to approximately 5 years)
Population: REP included all participants who received at least 1 dose of study drug and had a Baseline and at least 1 postbaseline disease assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Azacitidine 75 mg/m^2 | Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2
Number analyzed (Participants) | 53 | 55
percentage of participants | 45 | 51
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2; Test type: Superiority; p = 0.560, Cochran-Mantel-Haenszel — P-value is from an unstratified Cochran-Mantel Haenszel chi-square test; Absolute Rate Difference = 5.63, 95% CI 2-sided [-13.19 to 24.44] — [estimate comment as in outcome 6, analysis 1]

8. Secondary Outcome: Percentage of Participants With Overall Response
Description: Disease responses (HR MDS/CMML): modified IWG criteria for MDS; low-blast (LB) AML: revised IWG criteria for AML. Overall response(HR MDS/CMML)=CR,PR/HI,LB AML=CR+ CR with incomplete blood count recovery(Cri)+PR.HR MDS/CMML-CR:<=5%myeloblasts with normal maturation of bone marrow (BM) cell lines,>=11g/dL Hb,>=100*10^9/L plt,>=1.0*10^9/L ANC,0% blasts in peripheral blood; PR:CR criteria met except BM blasts>=50%less over pretreatment but still>5%; HI:hb increase (inc)>=1.5g/dL if baseline<11g/dL;plt inc>=30*10^9/L if baseline>20*10^9/L/Inc. from <20*10^9/L->20*10^9/L, ANC inc. by 100%;absolute inc. of>0.5*10^9/L if baseline<100*10^9/L. LB AML-CR:morphologic leukemia-freestate>1.0*10^9ANC,>=100*10^9/L plt, transfusion independence, no residual evidence of extramedullary leukemia;CRi:fulfill CR criteria except residual neutropenia<1.0*10^9/L/TTP<100*10^9/L;PR:all CR hematological values but>=50%less in BM aspirate. The percentages are rounded off to report the nearest whole numbers.
Time Frame: From date of randomization until CR, PR, or hematologic improvement (HI) (up to approximately 5 years)
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Azacitidine 75 mg/m^2 | Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2
Number analyzed (Participants) | 53 | 55
percentage of participants | 62 | 71
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2; Test type: Superiority; p = 0.343, Cochran-Mantel-Haenszel — P-value is from an unstratified Cochran-Mantel Haenszel chi-square test; Absolute Rate Difference = 8.64, 95% CI 2-sided [-9.09 to 26.38] — [estimate comment as in outcome 6, analysis 1]

9. Secondary Outcome: Percentage of Participants With CR in Low-blast AML
Description: Disease response for low-blast AML is based on the revised IWG response criteria for AML. CR for low-blast AML: morphologic leukemia-free state, ANC of more than 1.0*10^9/L and plt of >=1.0*10^9/L, transfusion independence, and no residual evidence of extramedullary leukemia. CR with incomplete blood count recovery for low-blast AML: some participants fulfill all of the criteria for CR except for residual neutropenia (<1.0*10^9/L) or thrombocytopenia (TTP) (<100*10^9/L). The percentages are rounded off to report the nearest whole numbers.
Time Frame: From date of randomization until CR (up to approximately 5 years)
Population: REP included all participants who received at least 1 dose of study drug and had a Baseline and at least 1 postbaseline disease assessment. Overall number analyzed are the number of participants with data available for analyses.
Measure: Number; unit: percentage of participants
Arm/Group | Azacitidine 75 mg/m^2 | Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2
Number analyzed (Participants) | 15 | 17
percentage of participants | 60.0 | 41.2
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2; Test type: Superiority; p = 0.296, Cochran-Mantel-Haenszel — P-value is from an unstratified Cochran-Mantel-Haenszel chi-square test; Absolute Rate Difference = -18.82, 95% CI 2-sided [-52.91 to 15.26] — [estimate comment as in outcome 6, analysis 1]

10. Secondary Outcome: Percentage of Participants With CR by Cycle 4
Description: Disease responses for HR MDS or CMML were based on modified IWG response criteria for MDS and for low-blast AML on revised IWG response criteria for AML. CR for HR MDS or CMML: <=5% myeloblasts with normal maturation of all cell lines in bone marrow, and >=11 g/dL Hb, >=100*10^9/L plt, ANC >=1.0*10^9/L and 0% blasts in peripheral blood. CR for low-blast AML: morphologic leukemia-free state, ANC of more than 1.0*10^9/L and plt of >=100*10^9/L, transfusion independence, no residual evidence of extramedullary leukemia. CR with incomplete blood count recovery for low-blast AML: some participants fulfill all criteria for CR except for residual neutropenia (<1.0*10^9/L)/TTP (<100*10^9/L). The percentages are rounded off to report the nearest whole numbers.
Time Frame: From date of randomization until CR by Cycle 4 (cycle length is equal to [=] 28 days)
Population: REP included all participants who received at least 1 dose of study drug and had a Baseline and at least 1 postbaseline disease assessment. Overall number analyzed is the number of participants with data available for analyses.
Measure: Number; unit: percentage of participants
Arm/Group | Azacitidine 75 mg/m^2 | Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2
Number analyzed (Participants) | 38 | 38
percentage of participants | 13.2 | 26.3
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2; Test type: Superiority; p = 0.152, Cochran-Mantel-Haenszel — P-value is from an unstratified Cochran-Mantel Haenszel chi-square test; Absolute Rate Difference = 13.16, 95% CI 2-sided [-4.49 to 30.81] — [estimate comment as in outcome 6, analysis 1]

11. Secondary Outcome: Percentage of Participants With CR and PR by Cycle 4
Description: Disease responses for HR MDS/CMML per modified IWG response criteria for MDS and for low-blast AML on revised IWG response criteria for AML.CR for HR MDS/CMML: <=5% myeloblasts with normal maturation of all cell lines in bone marrow, >=11 g/dL Hb; >=100*10^9/L plt; >=1.0*10^9/L ANC and 0% blasts in peripheral blood.PR for HR MDS/CMML: considered achieved if all CR criteria is met except for bone marrow blasts decreased by>=50% over pretreatment but still>5%.CR for low-blast AML: morphologic leukemia-free state, ANC of>1.0*10^9/L and plt of>=100*10^9/L, transfusion independence, no residual evidence of extramedullary leukemia. CR with incomplete blood count recovery for low-blast AML: fulfill all criteria for CR except for residual neutropenia (<100*10^9/L)/TTP (<100*10^9/L). PR for low-blast AML: all hematological values for CR but with decrease of >=50% in percentage of blasts to 5%-25% in bone marrow aspirate. The percentages are rounded off to report the nearest whole numbers.
Time Frame: From date of randomization until CR and PR, by Cycle 4 (cycle length=28 days)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Azacitidine 75 mg/m^2 | Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2
Number analyzed (Participants) | 38 | 38
percentage of participants | 21.1 | 31.6
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2; Test type: Superiority; p = 0.301, Cochran-Mantel-Haenszel — P-value is from an unstratified Cochran-Mantel Haenszel chi-square test; Absolute Rate Difference = 10.53, 95% CI 2-sided [-9.13 to 30.18] — [estimate comment as in outcome 6, analysis 1]

12. Secondary Outcome: Percentage of Participants With Overall Response by Cycle 4
Description: as for outcome 8
Time Frame: From date of randomization until CR, PR or HI, by Cycle 4 (cycle length=28 days)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Azacitidine 75 mg/m^2 | Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2
Number analyzed (Participants) | 38 | 38
percentage of participants | 44.7 | 57.9
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2; Test type: Superiority; p = 0.254, Cochran-Mantel-Haenszel — P-value is from an unstratified Cochran-Mantel Haenszel chi-square test; Absolute Rate Difference = 13.16, 95% CI 2-sided [-9.12 to 35.44] — [estimate comment as in outcome 6, analysis 1]

13. Secondary Outcome: Percentage of Participants With CR in Low-blast AML by Cycle 4
Description: Disease response for low-blast AML is based on revised IWG response criteria for AML. CR for low-blast AML: morphologic leukemia-free state, ANC of more than 1.0*10^9/L and ptl of >=100*10^9/L, transfusion independence, no residual evidence of extramedullary leukemia. CR with incomplete blood count recovery for low-blast AML: some participants fulfill all criteria for CR except for residual neutropenia (<1.0*10^9/L)/TTP (<100*10^9/L). The percentages are rounded off to report the nearest whole numbers.
Time Frame: From the date of randomization until CR by Cycle 4 (cycle length=28 days)
Population: REP included all participants who received at least 1 dose of study drug and had a Baseline and at least 1 postbaseline disease assessment. Data is reported for low blast AML participants which is included as the overall number of participants analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Azacitidine 75 mg/m^2 | Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2
Number analyzed (Participants) | 15 | 17
percentage of participants | 40.0 | 35.3
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2; Test type: Superiority; p = 0.787, Cochran-Mantel-Haenszel — P-value is from an unstratified Cochran-Mantel Haenszel chi-square test; Absolute Rate Difference = -4.71, 95% CI 2-sided [-38.33 to 28.92] — [estimate comment as in outcome 6, analysis 1]

14. Secondary Outcome: Duration of Complete Remission (CR)
Description: Duration of CR is first documented CR to the first documentation of PD or relapse from CR (participants with low-blast AML) or relapse after CR or PR (participants with HR MDS/CMML). Disease responses for HR MDS or CMML are based on the Modified IWG Response Criteria for MDS and for low-blast AML on the Revised IWG Response Criteria for AML.CR for HR MDS or CMML≤5% myeloblasts with normal maturation of all cell lines in the bone marrow,≥11 g/dL Hgb,≥100*10^9/L pl,≥1.0*10^9/L neutrophils;0% blasts in peripheral blood.CR for low-blast AML:morphologic leukemia-free state,neutrophils of<1.0*10^9/L;pl of≥100*10^9/L,transfusion independence,no residual evidence of extramedullary leukemia.CRi for low-blast AML: participants fulfill all of the criteria for CR except for residual neutropenia (<1.0*10^9/L) or thrombocytopenia (pl<100*10^9/L).
Time Frame: From date of randomization until CR (up to approximately 5 years)
Population: REP included all participants who received at least 1 dose of study drug and had a Baseline and at least 1 postbaseline disease assessment. Data is reported for the responders with complete remission.
Measure: Median (Full Range); unit: months
Arm/Group | Azacitidine 75 mg/m^2 | Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2
Number analyzed (Participants) | 19 | 25
months | 12.9 [8.31 to NA] — The upper limit of full range was not estimable due to low number of participants with the event. | 18.6 [9.00 to NA] — The upper limit of full range was not estimable due to low number of participants with the event.
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2; Test type: Superiority; p = 0.620, Log Rank — P-value is from an unstratified log-rank test; Hazard Ratio (HR) = 0.789, 95% CI 2-sided [0.308 to 2.020] — Hazard ratio was based on an unstratified Cox proportional hazard regression model and treatment as a factor in the model

15. Secondary Outcome: Duration of Complete Remission (CR) and Partial Remission (PR)
Description: Duration of CR is first documented CR to the first documentation of PD or relapse from CR (participants with low-blast AML). Disease responses (HR MDS/CMML) are based on modified IWG response criteria for MDS and for low-blast AML on revised IWG response criteria for AML. For HR MDS/CMML-CR:<=5%myeloblasts with normal maturation of all bone marrow cell lines, >=11 g/dL Hb, >=100*10^9/L plt,>=1.0*10^9/L neutrophils, 0% blasts in peripheral blood;PR: all CR criteria met except bone marrow blasts >=50% decrease over pretreatment but still >5%; low-blast AML-CR: morphologic leukemia-free state, >1.0*10^9/L ANC ,plt >=100*10^9/L,transfusion independence, no residual evidence of extramedullary leukemia;CR with incomplete blood count recovery:fulfill CR criteria except residual neutropenia <1.0*10^9/L/TTP <100*10^9/L;PR:all CR hematological values but with a decrease of >=50% in blasts percentage to 5%-25% in bone marrow aspirate.
Time Frame: From date of randomization until CR or PR (up to approximately 5 years)
Population: REP included all participants who received at least 1 dose of study drug and had a Baseline and at least 1 postbaseline disease assessment. Data is reported for the responders with complete CR and PR.
Measure: Median (Full Range); unit: months
Arm/Group | Azacitidine 75 mg/m^2 | Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2
Number analyzed (Participants) | 24 | 28
months | 12.9 [8.31 to NA] — The upper limit of 95% CI was not estimable due to low number of participants with the event. | 18.6 [10.15 to NA] — The upper limit of 95% CI was not estimable due to low number of participants with the event.
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2; Test type: Superiority; p = 0.436, Log Rank — P-value is from an unstratified log-rank test; Hazard Ratio (HR) = 0.719, 95% CI 2-sided [0.313 to 1.653] — [estimate comment as in outcome 14, analysis 1]

16. Secondary Outcome: Duration of Overall Response
Description: Duration of OR: response to first documentation of PD or relapse from CR for low-blast AML or relapse after CR or PR for HR MDS/CMML. Disease responses(HR MDS/CMML): modified IWG criteria for MDS;low-blast AML: revised IWG criteria for AML.Overall response(HR MDS/CMML)=CR,PR/HI,LB AML=CR+ Cri+PR.HR MDS/CMML-CR:≤5%myeloblasts with normal maturation of BM cell lines,≥11g/dL Hb,≥100*10^9/L plt,≥1.0*10^9/L ANC,0%blasts in peripheral blood; PR:CR criteria met except BM blasts≥50%less over pretreatment but still>5%; HI:hb increase(inc)≥1.5g/dL if baseline<11g/dL; plt inc≥30*10^9/L if baseline >20*10^9/L inc from<20*10^9/L->20*10^9/L,ANC inc by100%; absolute inc of >0.5*10^9/L if baseline <100*10^9/L.LB AML-CR: morphologic leukemia-freestate >1.0*10^9 ANC,≥100*1 ^9/Lplt, transfusion independence, no residual evidence of extramedullary leukemia; CRi:fulfill CR criteria except residual neutropenia<1.0*10^9/L/TTP<100*10^9/L; PR:all CR hematological values but>=50%less in BM aspirate.
Time Frame: From date of randomization until CR, PR or HI (up to approximately 5 years)
Population: REP included all participants who received at least 1 dose of study drug and had a Baseline and at least 1 postbaseline disease assessment. Data is reported for overall responders.
Measure: Median (Full Range); unit: months
Arm/Group | Azacitidine 75 mg/m^2 | Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2
Number analyzed (Participants) | 33 | 39
months | 14.0 [12.62 to NA] — The upper limit of full range was not estimable due to lower number of participants with the event. | 20.6 [10.71 to NA] — The upper limit of full range was not estimable due to lower number of participants with the event.
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2; Test type: Superiority; p = 0.565, Log Rank — P-value is from an unstratified log-rank test; Hazard Ratio (HR) = 0.810, 95% CI 2-sided [0.395 to 1.662] — [estimate comment as in outcome 14, analysis 1]

17. Secondary Outcome: Duration of Complete Remission (CR) in Low-blast AML
Description: Disease responses for low-blast AML is based on revised IWG response criteria for AML. CR for low-blast AML: morphologic leukemia-free state, ANC of more than 1.0*10^9/L and plt of >=100*10^9/L, transfusion independence, no residual evidence of extramedullary leukemia. CR with incomplete blood count recovery for low-blast AML: some participants fulfill all criteria for CR except for residual neutropenia (<1.0*10^9/L)/TTP (<100*10^9/L).
Time Frame: From date of randomization until CR (up to approximately 5 years)
Population: REP included all participants who received at least 1 dose of study drug and had a Baseline and at least 1 postbaseline disease assessment. Data is reported for responders with low blast AML having complete remission.
Measure: Median (Full Range); unit: months
Arm/Group | Azacitidine 75 mg/m^2 | Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2
Number analyzed (Participants) | 4 | 4
months | 10.2 [0.2 to 10.2] | 12.6 [5.6 to 44.0]
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2; Test type: Superiority; p = 0.383, Log Rank — P-value comparing duration of CR in low blast AML between treatment groups is based on unstratified log-rank test; Hazard Ratio (HR) = 0.420, 95% CI 2-sided [0.057 to 3.109] — [estimate comment as in outcome 14, analysis 1]

18. Secondary Outcome: Time to First CR or PR
Description: Time to first CR or PR: time from randomization to first documented CR or PR, whichever occurs first. Disease responses (HR MDS/CMML) based on modified IWG response criteria for MDS; low-blast AML on revised IWG response criteria for AML. HR MDS/CMML-CR: <=5% myeloblasts with normal maturation of all bone marrow cell lines, >=11 g/dL Hb, >=100*10^9/L plt,>=1.0*10^9/L ANC, 0% blasts in peripheral blood; PR: all CR criteria met except bone marrow blasts >=50% decrease over pretreatment but still >5%; For low-blast AML-CR: morphologic leukemia-free state, >1.0*10^9/L ANC, plt >=100*10^9/L, transfusion independence, no residual evidence of extramedullary leukemia; CR with incomplete blood count recovery: fulfill CR criteria except residual neutropenia <1.0*10^9/L/TTP <100*10^9/L; PR: all CR hematological values but with a decrease of >=50% in the percentage of blasts to 5% to 25% in the bone marrow aspirate.
Time Frame: From date of randomization until CR or PR (up to approximately 5 years)
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Azacitidine 75 mg/m^2 | Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2
Number analyzed (Participants) | 53 | 55
months | 13.2 [6.4 to NA] — The upper limit of 95% CI was not estimable due to low number of participants with the event. | 8.3 [4.5 to NA] — The upper limit of 95% CI was not estimable due to low number of participants with the event.
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2; Test type: Superiority; p = 0.498, Log Rank — P-value is from an unstratified log-rank test; Hazard Ratio (HR) = 1.206, 95% CI 2-sided [0.699 to 2.081] — HR is based on an unstratified Cox proportional hazard regression model with treatment as a factor. HR>1 for the treatment indicates a shorter time to first CR, CRi or PR in the Pevonedistat Combination arm compared to the Azacitidine only arm

19. Secondary Outcome: Time to Subsequent Therapy
Description: Time to subsequent therapy is defined as time from randomization to the date of the first subsequent therapy. Subsequent therapy is defined as agent(s) with antileukemic/anti-MDS activity. Participants who discontinue study treatment to receive single-agent azacitidine off study did not be counted as receiving subsequent therapy.
Time Frame: From date of randomization up to approximately 5 years
Population: ITT Population was defined as all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Azacitidine 75 mg/m^2 | Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2
Number analyzed (Participants) | 62 | 58
months | NA [NA to NA] — The median and 95% CI was not estimable due to low number of participants with the event. | NA [NA to NA] — The median and 95% CI was not estimable due to lower number of participants with the event.
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2; Test type: Superiority; p = 0.888, Log Rank — P-value is from an unstratified log-rank test; Hazard Ratio (HR) = 0.905, 95% CI 2-sided [0.226 to 3.620] — HR is based on an unstratified Cox proportional hazard regression model with treatment as a factor. HR<1for the treatment indicates a longer time to Subsequent Therapy in the Pevonedistat Combination arm compared to the Azacitidine only arm

20. Secondary Outcome: Percentage of Participants With Red Blood Cells (RBCs) and Platelet-transfusion Independence
Description: A participant was defined as RBC or platelet-transfusion independent if he/she received no RBC or platelet transfusions for a period of at least 8 weeks before the first dose of study drug through 30 days after the last dose of any study drug. Rate of transfusion independence was defined as number of participants who became transfusion independent divided by the number of participants who were transfusion dependent at Baseline.
Time Frame: 8 weeks before randomization through 30 days after last dose of any study drug (up to approximately 5 years and 3 months)
Population: ITT Population included all participants who were randomized. Overall number analyzed are the number of participants from a subset of the ITT Population who were transfusion dependent at Baseline. Number analyzed is the number of participants who were transfusion dependent at Baseline for the specified category.
Measure: Number; unit: percentage of participants
Arm/Group | Azacitidine 75 mg/m^2 | Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2
Number analyzed (Participants) | 26 | 26
percentage of participants
  RBCs-transfusion Independence | 50.0 | 69.2
  Platelet-transfusion Independence: number analyzed (Participants) | 10 | 5
  Platelet-transfusion Independence | 60.0 | 80.0
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2; Percentage of Participants With RBCs-transfusion Independence; Test type: Superiority; p = 0.162, Cochran-Mantel-Haenszel — P-value is from an unstratified Cochran-Mantel Haenszel chi-square test; Absolute Rate Difference = 19.231, 95% CI 2-sided [-6.925 to 45.386]
Statistical Analysis 2: Comparison: Azacitidine 75 mg/m^2 vs Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2; Percentage of Participants With Platelet-transfusion Independence; Test type: Superiority; p = 0.454, Cochran-Mantel-Haenszel — P-value is from an unstratified Cochran-Mantel Haenszel chi-square test; Absolute Rate Difference = 20.000, 95% CI 2-sided [-26.381 to 66.381]

21. Secondary Outcome: Percentage of Participants With at Least 1 Inpatient Hospital Admissions Related to HR MDS, CMML or Low-blast AML
Description: Inpatient hospital admission data was collected through transformation to AML (HR MDS/CMML participants) or disease progression (low-blast AML participants) or until initiation of subsequent therapy (all participants), whichever occurred first. Transformation to AML is defined, according to WHO Classification, as a participant having 20% blasts in the blood or marrow and increase of blast count by 50%. Percentage of participants was calculated as the total number of events divided by the total number of subject-years in each group.
Time Frame: From date of randomization until transformation to AML or until initiation of subsequent therapy (up to approximately 5 years)
Population: ITT Population included all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Azacitidine 75 mg/m^2 | Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2
Number analyzed (Participants) | 62 | 58
percentage of participants | 0.4811 [0.37956 to 0.58265] | 0.5878 [0.42606 to 0.74953]

22. Secondary Outcome: Time to Progressive Disease (PD), Relapse, or Death
Description: Time from randomization until PD/transformation to AML/relapse/death due to any cause, whichever occurs first. Relapse after CR or PR in MDS/CMML: return to pretreatment bone marrow blast % or decrement of >=50% from maximum remission levels in ANC or plt, reduction in Hb concentration by >=1.5 g/dL or transfusion dependence. PD: at least 50% decrement from maximum remission in ANC or plt, or reduction in Hb by>=2g/dL or transfusion dependence;participants with <5% blasts: >=50% increase (inc) in blasts to >5%; 5%-10%: >=50% inc to >10%; 10%-20%: >=50% inc to>20%;20%-30%:>=50% inc to >30%. Relapse after CR in Low blast AML: reappearance of leukemic blasts in peripheral blood or >=5% blasts in bone marrow not attributable to any cause (example, bone marrow regeneration after consolidation therapy). If there are no circulating blasts, bone marrow contains 5%-20% blasts, a repeat analysis is performed a week later.
Time Frame: From date of randomization until PD, relapse or death (up to approximately 5 years)
Population: ITT Population was defined as all participants who were randomized.
Measure: Median (Full Range); unit: months
Arm/Group | Azacitidine 75 mg/m^2 | Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2
Number analyzed (Participants) | 62 | 58
months | 13.6 [9.40 to 16.53] | 15.2 [12.39 to 20.83]
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2; Test type: Superiority; p = 0.266, Log Rank — P-value is from an unstratified log-rank test; Hazard Ratio (HR) = 0.790, 95% CI 2-sided [0.521 to 1.198] — HR is based on an unstratified Cox proportional hazard regression model with treatment as a factor. HR<1for the treatment indicates a longer time to PD, Relapse, or Death in the Pevonedistat Combination arm compared to the Azacitidine only arm

23. Secondary Outcome: Number of Participants Reporting One or More Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. A SAE was defined as any untoward medical occurrence that: 1) results in death, 2) is life-threatening, 3) requires inpatient hospitalization or prolongation of existing hospitalization, 4) results in persistent or significant disability/incapacity, 5) leads to a congenital anomaly/birth defect in the offspring of the participant or 6) is an medically important event that satisfies any of the following: a) May require intervention to prevent items 1 through 5 above. b) May expose the participant to danger, even though the event is not immediately life threatening or fatal or does not result in hospitalization. A TEAE was defined as any adverse event occurring after the start of pevonedistat administration of the treatment period.
Time Frame: From date of first dose up to 30 days after administration of the last dose of any study drug (up to approximately 5 years)
Population: Safety Population included all enrolled participants who receive at least 1 dose of any study drug azacitidine alone or pevonedistat + azacitidine.
Measure: Count of Participants; unit: Participants
Groups:
- Azacitidine 75 mg/m^2: Azacitidine 75 milligram per square meter (mg/m^2), infusion, intravenously or subcutaneously, on Days 1 to 5, and on Days 8 and 9 in 28-day treatment cycles until unacceptable toxicity, relapse, transformation to AML (for participants with HR MDS or CMML), or progressive disease (for participants with low-blast AML).
- Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2: Azacitidine 75 mg/m^2, infusion, intravenously or subcutaneously, on Days 1 to 5, and on Days 8 and 9 and pevonedistat 20 mg/m^2, infusion, intravenously, on Days 1, 3, and 5 in 28-day treatment cycles until unacceptable toxicity, relapse, transformation to AML (for participants with HR MDS or CMML), or progressive disease (for participants with low-blast AML).
Arm/Group | Azacitidine 75 mg/m^2 | Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2
Number analyzed (Participants) | 62 | 58
Participants
  TEAEs | 62 | 57
  SAEs | 40 | 40

24. Secondary Outcome: Number of Participants in the Safety Analysis Population With Clinically Significant Laboratory Abnormalities Reported as TEAEs
Description: Laboratory assessments included clinical chemistry, hematology, and urinalysis.
Time Frame: as for outcome 23
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Azacitidine 75 mg/m^2 | Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2
Number analyzed (Participants) | 62 | 58
Participants
  Neutropenia | 21 | 21
  Anaemia | 29 | 19
  Neutrophil count decreased | 6 | 12
  Thrombocytopenia | 15 | 16

25. Secondary Outcome: Number of Participants With Change From Baseline Values in Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: Number of participants with change from Baseline in ECOG performance status was measured on 6 point scale to assess participant's performance status, where: Grade 0(Normal activity. Fully active, able to carry on all pre-disease activities without restriction); Grade 1(Symptoms but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to carry out light or sedentary work); Grade 2(In bed <50% of the time. Ambulatory and capable of all self-care, but unable to carry out any work activities. Up and about more than 50% of waking hours); Grade 3(In bed >50% of the time. Capable of only limited self-care, confined to bed or chair more than 50 percent of waking hours); Grade 4(100% bedridden. Completely disabled, cannot carry on any self-care, totally confined to bed or chair); Grade 5(Dead).
Time Frame: as for outcome 23
Population: ITT population was defined as all participants who were randomized in the Safety Population. Only categories for which there was at least 1 participant are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Azacitidine 75 mg/m^2 | Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2
Number analyzed (Participants) | 62 | 58
Participants
  Baseline: 0; Overall: 0 | 13 | 9
  Baseline: 0; Overall: 1 | 15 | 13
  Baseline: 0; Overall: 2 | 3 | 3
  Baseline: 0; Overall: 3 | 0 | 2
  Baseline: 0; Overall: 4 | 2 | 0
  Baseline: 1; Overall: 1 | 17 | 18
  Baseline: 1; Overall: 2 | 5 | 8
  Baseline: 1; Overall: 3 | 5 | 2
  Baseline: 2; Overall: 2 | 2 | 3

26. Secondary Outcome: Number of Participants in the Safety Analysis Population With Clinically Significant Change From Baseline in Electrocardiogram (ECG) Values Reported as TEAEs
Description: ECG assessments included QT, QRS duration, PR interval, ventricular rate, QTcB, QTcF.
Time Frame: as for outcome 23
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Azacitidine 75 mg/m^2 | Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2
Number analyzed (Participants) | 62 | 58
Participants
  Atrial fibrillation | 4 | 4
  Tachycardia | 1 | 4

27. Secondary Outcome: Number of Participants in the Safety Analysis Population With Clinically Significant Change From Baseline Values in Vital Signs Reported as TEAEs
Description: Vital signs assessments included diastolic and systolic blood pressure, heart rate, and body temperature.
Time Frame: as for outcome 23
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Azacitidine 75 mg/m^2 | Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2
Number analyzed (Participants) | 62 | 58
Participants
  Pyrexia | 25 | 22
  Hypotension | 3 | 6

ADVERSE EVENTS:
Time Frame: From first dose up to 30 days after administration of the last dose of any study drug (up to approximately 5 years)
Description: At each visit the investigator had to document any occurrence of adverse events, abnormal laboratory findings, and vital signs. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Azacitidine 75 mg/m^2 | Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2
All-Cause Mortality (participants affected / at risk) | 50/62 | 47/58
Serious Adverse Events (participants affected / at risk) | 40/62 | 40/58
Other Adverse Events (participants affected / at risk) | 58/62 | 51/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azacitidine 75 mg/m^2 (N=62) | Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2 (N=58)
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Abscess limb (Infections and infestations) | 0 | 1
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Anuria (Renal and urinary disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1
Arthritis infective (Infections and infestations) | 0 | 1
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Bacteraemia (Infections and infestations) | 1 | 2
Bacterial sepsis (Infections and infestations) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cauda equina syndrome (Nervous system disorders) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 2
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Coronavirus infection (Infections and infestations) | 0 | 1
Death (General disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Drug hypersensitivity (Immune system disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Embolic stroke (Nervous system disorders) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 2
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 15 | 13
Gastric haemorrhage (Gastrointestinal disorders) | 2 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal ulcer perforation (Gastrointestinal disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hepatic lesion (Hepatobiliary disorders) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Influenza (Infections and infestations) | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Ischaemic gastritis (Gastrointestinal disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 2
Multiple organ dysfunction syndrome (General disorders) | 1 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome transformation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Oral viral infection (Infections and infestations) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Parophthalmia (Eye disorders) | 0 | 1
Peripheral venous disease (Vascular disorders) | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 7 | 8
Post procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0
Proctitis (Gastrointestinal disorders) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 1
Pyrexia (General disorders) | 6 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
SARS-CoV-2 test positive (Investigations) | 0 | 1
Sepsis (Infections and infestations) | 4 | 4
Sinusitis (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 0
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 1
Viral infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azacitidine 75 mg/m^2 (N=62) | Azacitidine 75 mg/m^2 + Pevonedistat 20 mg/m^2 (N=58)
Abdominal pain (Gastrointestinal disorders) | 10 | 3
Acute kidney injury (Renal and urinary disorders) | 0 | 4
Alanine aminotransferase increased (Investigations) | 4 | 4
Anaemia (Blood and lymphatic system disorders) | 27 | 19
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 6
Aspartate aminotransferase increased (Investigations) | 5 | 4
Asthenia (General disorders) | 13 | 18
Atrial fibrillation (Cardiac disorders) | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 9
Blood alkaline phosphatase increased (Investigations) | 0 | 3
Blood bilirubin increased (Investigations) | 0 | 3
Blood creatinine increased (Investigations) | 0 | 3
Bronchitis (Infections and infestations) | 7 | 0
Chills (General disorders) | 7 | 4
Conjunctival haemorrhage (Eye disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 29 | 21
Contusion (Injury, poisoning and procedural complications) | 4 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 22
Decreased appetite (Metabolism and nutrition disorders) | 13 | 11
Dehydration (Metabolism and nutrition disorders) | 4 | 0
Depression (Psychiatric disorders) | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 17 | 19
Dizziness (Nervous system disorders) | 9 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 13
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Dysuria (Renal and urinary disorders) | 0 | 4
Ear pain (Ear and labyrinth disorders) | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 13
Erythema (Skin and subcutaneous tissue disorders) | 5 | 4
Fall (Injury, poisoning and procedural complications) | 6 | 8
Fatigue (General disorders) | 25 | 12
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 0
Haematoma (Vascular disorders) | 0 | 7
Haematuria (Renal and urinary disorders) | 0 | 3
Haemorrhoids (Gastrointestinal disorders) | 0 | 5
Headache (Nervous system disorders) | 8 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 4
Hypertension (Vascular disorders) | 0 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 0
Hypotension (Vascular disorders) | 0 | 6
Injection site pain (General disorders) | 7 | 4
Injection site reaction (General disorders) | 0 | 3
Insomnia (Psychiatric disorders) | 7 | 6
Malaise (General disorders) | 4 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Nasopharyngitis (Infections and infestations) | 4 | 7
Nausea (Gastrointestinal disorders) | 28 | 21
Neutropenia (Blood and lymphatic system disorders) | 21 | 21
Neutrophil count decreased (Investigations) | 6 | 12
Non-cardiac chest pain (General disorders) | 4 | 0
Oedema peripheral (General disorders) | 9 | 12
Oral candidiasis (Infections and infestations) | 4 | 3
Oral herpes (Infections and infestations) | 6 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Pain (General disorders) | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 10
Pallor (Vascular disorders) | 0 | 3
Peripheral swelling (General disorders) | 0 | 5
Petechiae (Skin and subcutaneous tissue disorders) | 4 | 0
Platelet count decreased (Investigations) | 7 | 7
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Pneumonia (Infections and infestations) | 8 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 3
Pyrexia (General disorders) | 22 | 21
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 3
Respiratory tract infection (Infections and infestations) | 0 | 3
Somnolence (Nervous system disorders) | 0 | 3
Stomatitis (Gastrointestinal disorders) | 5 | 0
Tachycardia (Cardiac disorders) | 0 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 15 | 15
Urinary tract infection (Infections and infestations) | 5 | 5
Vomiting (Gastrointestinal disorders) | 13 | 14
Weight decreased (Investigations) | 5 | 5
White blood cell count decreased (Investigations) | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-07-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT02610777/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/77/NCT02610777/SAP_001.pdf